CLINICAL TRIAL: NCT04968665
Title: The Mechanism for the Effects of Joint Biomechanical Properties on Medial Cartilage of Tibiofemoral Joint Degeneration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Ren Shuang, associate researcher, Peking University Third Hospital
Other Study IDs: M2019434
Record Dates: First submitted 2021-07-02; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Anterior Cruciate Ligament Injuries; Cartilage Degeneration
Keywords: sports biomechanics; joint loading; anterior cruciate ligament reconstruction; cartilage degeneration; functional MRI
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: gait testing and MRI at baseline for healthy volunteers
  Interventions: Diagnostic Test: gait testing, functional MRI
- ACL-deficient patients: gait testing and MRI at pre-operation, 6 months post-operation, 1 year post-operation, 2 years post-operation
  Interventions: Diagnostic Test: gait testing, functional MRI

INTERVENTIONS:
Diagnostic Test: gait testing, functional MRI — diagnostic tests including the gait testing and functional MRI

SUMMARY:
Explore The Mechanism for the Effects of Joint Biomechanical Properties on Medial Cartilage of Tibiofemoral Joint Degeneration

DETAILED DESCRIPTION:
Cartilage degeneration in the medial tibiofemoral joint is common after anterior cruciate ligament reconstruction (ACLR), which may develop into knee osteoarthritis (disability rate 21.3%). Alterations in joint biomechanical properties play an important role in cartilage degeneration after ACLR. However, the mechanism remains unclear.

Our research studied the joint kinematics and kinetics properties after ACLR and found significant changes in biomechanics in the ACLR knees. Therefore, this study will combine longitude biochemical changes in the cartilage to explore how the alterations in biomechanics would influence biochemical changes in the joint cartilage.

This study will explore the joint biomechanical properties during functional activities by motion analysis, the effects of biomechanical properties on cartilage stress distribution by finite element analysis, the long-term biochemical changes in the joint cartilage by functional MRI. This study will establish prediction models for cartilage biomechanical changes in the mid-term based on joint biomechanical properties in the early stage after ACLR, and cartilage biomechanical changes in the long-term based on joint biomechanical properties in the mid-term after ACLR. The study aims to clarify the mechanism of cartilage degeneration after ACLR and search biomechanical risk factors, in order to provide methods for clinical prevention of cartilage degeneration after ACLR.

ELIGIBILITY:
Inclusion Criteria:

Unilateral ACL rupture of the knee

Exclusion Criteria:

concomitant with other ligament injury or rupture, with history of surgery or musculoskeletal system injury of the contralateral knee, and the time from injury to operation more than 8 weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Thirty patients with ACL rupture undergoing ACL reconstruction surgery at the Institute of Sports Medicine, Peking University Third Hospital would be included in the study cohort were included, A total of 30 healthy volunteers with no history of musculoskeletal system injury or surgery in bilateral lower extremities would be included
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
knee T1 rho value | On the day of enrollment.
  knee T1 rho value by functional MRI
knee T1 rho value | At 6 months post operation.
  knee T1 rho value by functional MRI
knee T1 rho value | At 12 months post operation.
  knee T1 rho value by functional MRI
knee T1 rho value | At 2 years post operation.
  knee T1 rho value by functional MRI
knee T2 value | On the day of enrollment.
  knee T1 rho value by functional MRI
knee T2 value | At 6 months post operation.
  knee T1 rho value by functional MRI
knee T2 value | At 12 months post operation.
  knee T1 rho value by functional MRI
knee T2 value | At 2 years post operation.
  knee T1 rho value by functional MRI
knee extension angles | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee extension angles | At 6 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee extension angles | At 12 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee extension angles | At 2 years post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee moments | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee moments | At 6 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee moments | At 12 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee moments | At 2 years post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
ground reaction force | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
ground reaction force | At 6 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
ground reaction force | At 12 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
ground reaction force | At 2 years post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee rotation angles | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee rotation angles | At 6 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee rotation angles | At 12 months post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping
knee rotation angles | At 2 years post operation.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Ren, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No